CLINICAL TRIAL: NCT03847987
Title: A 2 Part, Randomized, Open-Label, Single Dose, Crossover Study to Assess the Relative Bioavailability of Phase II Tablet Formulation Compared to the Current Phase I Capsule Formulation and the Effect of Food and Taste Assessment on the Phase II Tablet Formulation in Healthy Participants
Brief Title: A 2 Part Study to Assess the Relative Bioavailability of Tablet Formulation Compared to Capsule Formulation and the Effect of Food and Taste Assessment on the Tablet Formulation in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BP40950
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Results first posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Flavoring Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Participants will receive 4 single oral doses of RO7017773 under either fed or fasted conditions, one of which will be a taste assessment. There will be a 7-10 day washout period between doses.
  Interventions: Drug: RO7017773 Phase I Capsule; Drug: RO7017773 Phase II Tablet Unflavored
- Part 2 (Experimental): Participants will receive 2 single oral doses of RO7017773, either sweetened/flavored, or unflavored and dispersed in juice. There will be a 7-10 day washout period between doses.
  Interventions: Drug: RO7017773 Phase II Tablet Unflavored; Drug: RO7017773 Phase II Tablet Sweetened/Flavored

INTERVENTIONS:
Drug: RO7017773 Phase I Capsule — Participants will receive 1 single oral dose of RO7017773 Phase I Capsule.
  Arms: Part 1
Drug: RO7017773 Phase II Tablet Unflavored — Participants will receive 3 single oral doses of unflavored RO7017773 Phase II tablet during Part 1, and 1 single oral dose of unflavored RO7017773 Phase II tablet during Part 2.
Drug: RO7017773 Phase II Tablet Sweetened/Flavored — Participants will receive 1 single oral dose of sweetened/flavored RO7017773 Phase II tablet during Part 2.
  Arms: Part 2

SUMMARY:
This is a two-part, open-label, healthy volunteer study. Part I will investigate the relative bioavailability of capsule and tablet formulations of RO7017773. Part II will explore how the taste of the tablet formulation is perceived with and without added sweetener/flavoring.

ELIGIBILITY:
Inclusion Criteria

* Non-smoker for at least six months
* Healthy, as judged by the Investigator
* Women of non-childbearing potential (WONCBP) who are not pregnant or lactating
* Men must be willing to remain abstinent or agree to use contraceptive measures with partners who are women of childbearing potential (WOCBP), and must refrain from donating sperm, for at least 28 days after the last dose of study drug

Exclusion Criteria

* History or evidence of any medical condition potentially altering the absorption, metabolism or elimination of drugs
* History of convulsions (other than benign febrile convulsions of childhood) including epilepsy, or personal history of significant cerebral trauma or CNS infections (e.g. meningitis)
* A history of clinically significant hypersensitivity (e.g., drugs, excipients) or allergic reactions
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Have used or intend to use over-the-counter or prescription medication including herbal medications within 30 days prior to dosing
* Participation in an investigational drug or device study within 90 days prior to screening
* Human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening or within 3 months prior to starting study treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy male and female participants between ages 18-55 years, who were nonsmokers for at least 6 months.
Groups:
- Part 1: Sixteen (16) total participants received each of the following treatments, with a 7-10 day washout period between treatments:
  * Treatment A = A single oral dose of RO7017773 (capsule) swallowed whole under fasted conditions
  * Treatment B = A single oral dose of RO7017773 (tablet) swallowed whole under fasted conditions
  * Treatment C = A single oral dose of RO7017773 (tablet) swallowed whole under fed conditions
  * Treatment D = A single oral dose of RO7017773 (tablet) dispersed in water under fasted conditions
  Treatment sequences were randomly assigned
- Part 2: Eight (8) total participants received each of the following treatments, with a 7-10 day washout period between treatments:
  * Treatment A (taste assessment) = A single oral dose of RO7017773 (tablet) containing flavor/sweetener dispersed in water under fasted conditions
  * Treatment B (taste assessment) = A single oral dose of RO7017773 (tablet) with no flavor/sweetener dispersed in apple juice under fasted conditions
  Treatment sequences were randomly assigned
Period: Overall Study
Arm/Group | Part 1 | Part 2
Started | 16 | 8
Completed | 13 | 8
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 | Part 2 | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.1 (9.66) | 35.3 (10.57) | 33.7 (4.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 16 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 12 | 8 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of RO7017773 (Part 1)
Time Frame: Day 1 to Day 5
Population: The PK population included all participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 1 - Treatment A: Participants received a single oral dose of RO7017773 (capsule) swallowed whole under fasted conditions
- Part 1 - Treatment B: Participants received a single oral dose of RO7017773 (tablet) swallowed whole under fasted conditions
- Part 1 - Treatment C: Participants received a single oral dose of RO7017773 (tablet) swallowed whole under fed conditions
- Part 1 - Treatment D: Participants received a single oral dose of RO7017773 (tablet) dispersed in water under fasted conditions
Arm/Group | Part 1 - Treatment A | Part 1 - Treatment B | Part 1 - Treatment C | Part 1 - Treatment D
Number analyzed (Participants) | 16 | 16 | 16 | 16
ng/mL | 1320 (25.8) | 1570 (27.4) | 1120 (25.3) | 1490 (26.6)

2. Secondary Outcome: Taste Assessment, as Measured by Taste Questionnaire (Part 1)
Description: Taste was assessed using a questionnaire that asking participants to rate the overall taste of study drug dispersed in various vehicles on a scale from 1-5, with 1=no taste, and 5=very intense taste.
Time Frame: Day 1
Population: The population for this taste assessment was Part 1 - Treatment D (study drug dispersed in water).
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Part 1 - Treatment D
Number analyzed (Participants) | 14
Units on a Scale | 2 [1 to 3]

3. Primary Outcome: Cmax of RO7017773 (Part 2)
Time Frame: Day 1 to Day 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part 2 - Treatment A: Participants received a single oral dose of RO7017773 (tablet) containing flavor/sweetener dispersed in water under fasted conditions
- Part 2 - Treatment B: Participants received a single oral dose of RO7017773 (tablet) with no flavor/sweetener dispersed in apple juice under fasted conditions
Arm/Group | Part 2 - Treatment A | Part 2 - Treatment B
Number analyzed (Participants) | 8 | 8
ng/mL | 1470 (25.2) | 1210 (19.0)

4. Primary Outcome: Taste Assessment, as Measured by Taste Questionnaire (Part 2)
Description: as for outcome 2
Time Frame: Day 1
Population: The populations for this taste assessment were Part 2 - Treatment A and Part 2 - Treatment B.
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Part 2 - Treatment A | Part 2 - Treatment B
Number analyzed (Participants) | 8 | 8
Units on a Scale | 3 [1 to 4] | 1.5 [1 to 4]

5. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Baseline through end of study (approximately 6 weeks)
Measure: Number; unit: Percentage of Participants
Arm/Group | Part 1 - Treatment A | Part 1 - Treatment B | Part 1 - Treatment C | Part 1 - Treatment D | Part 2 - Treatment A | Part 2 - Treatment B
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 8 | 8
Percentage of Participants | 56.3 | 60.0 | 53.3 | 28.6 | 75.0 | 62.5

ADVERSE EVENTS:
Time Frame: Baseline through end of study (up to approximately 6 weeks)
Arm/Group | Part 1 - Treatment A | Part 1 - Treatment B | Part 1 - Treatment C | Part 1 - Treatment D | Part 2 - Treatment A | Part 2 - Treatment B
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/14 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/14 | 0/14 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 9/16 | 9/15 | 8/15 | 4/14 | 6/8 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1 - Treatment A (N=16) | Part 1 - Treatment B (N=15) | Part 1 - Treatment C (N=15) | Part 1 - Treatment D (N=14) | Part 2 - Treatment A (N=8) | Part 2 - Treatment B (N=8)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 3/14 (3) | 1 (1) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT03847987/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT03847987/SAP_001.pdf